CLINICAL TRIAL: NCT06763861
Title: SFINX - Sacral Neuromodulation and Faecal Incontinence and Its Unknown Effect on the External Anal Sphincter
Brief Title: Sacral Neuromodulation and Faecal Incontinence and Its Unknown Effect on the External Anal Sphincter
Acronym: SFINX
Status: Recruiting | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: Dnr 2024-04527-01
Record Dates: First submitted 2024-12-11; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Fecal Incontinence
Keywords: Fecal Incontinence; Sacral neuromodulation; Surgery; Pathology; Proctology; Quality of Life; Health status
MeSH Terms: conditions — Fecal Incontinence | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies from the external anal sphincter muscle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients without diagnosis of FI: Biopsies from EAS among patients diagnosed with rectal cancer and no records of previous diagnosis of FI and now receiving treatment with abdominoperineal resection.
  Interventions: Other: Biopsy
- Patients diagnosed with FI: Biopsies from EAS among patients diagnosed with FI and recieving treatment with sacral neuromodulation before implantation of the device and 12 months postoperatively.
  Interventions: Other: Biopsy

INTERVENTIONS:
Other: Biopsy — Biopsies from EAS

SUMMARY:
This innovative project aims to investigate structures and morphology of the external anal sphincter (EAS) as well as the impact of sacral neuromodulation (SNM) on the EAS morphology and biochemistry among patients with faecal incontinence (FI).

SNM is a well implemented treatment for FI and consist of electrical stimulation of sacral nerve roots to promote continence and may even contribute to total continence. It has shown a positive effects on both short- and long-term. The biologic effect of SNM on EAS is unknown.

The aim is to investigate the effect of SNM on EAS morphology, function, and biochemistry to help physicians and researchers to understand the underlying mechanisms of SNM and the anal sphincter complex to further improve and optimize treatment methods for patients with FI.

The research project consists of three phases. The first phase includes biopsies from the EAS among patients with no previous history of FI. These patients have been diagnosed with rectal cancer and will undergo surgery with abdominoperineal excision.

The second phase includes patients diagnosed with FI and subject for implantation of SNM for treatment of FI. Prior to implantation of SNM all patients will have been examined with 3D endo-anal ultrasound and anorectal manometry as well as answered questionnaires targeting general health, bowel dysfunction and FI. A biopsy of the superficial portion of the EAS is retrieved under local anaesthesia in connection to the test period for implantation of the SNM device.

The last phase, phase three, includes 3D endo-anal ultrasound, anorectal manometry, and a second biopsy of the EAS twelve months after implantation with SNM.

The histopathological analysis in all the three phases will include general morphology, distribution of cell nuclei, satellite cells, muscle fiber type, neural structures and connective tissue.

ELIGIBILITY:
Phase 1

Inclusion Criteria:

* ≥ 18 years of age
* Male or female
* Diagnosed with rectal cancer and receive treatment with abdominoperineal resection
* Signed an informed consent

Exclusion Criteria:

* Previous diagnosis of FI
* Unable to speak and/or read Swedish to ensure informed consent
* Tumour involving the sphincter complex or is in close connection

Phase 2 and 3

Inclusion Criteria:

* Diagnosed with FI and will receive treatment with sacral neuromodulation
* Male or female
* Signed an informed consent

Exclusion Criteria:

* Unable to speak and/or read Swedish to ensure informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Please see Study description.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The effect of sacral neuromodulation on the external anal sphincter muscle among patients with faecal incontinence | 2 years - The biopsies will be analysed and assessed continuously.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Strigård, Prof., Senior consultant, Study Chair — Department of Diagnostics and Interventions, Umeå University
Locations (1):
- Umeå University Hospital, Umeå, Västerbotten County, Sweden